CLINICAL TRIAL: NCT02058199
Title: A Pharmacodynamic Study of Rivaroxaban in Subjects Who Have Undergone Roux-en-Y Gastric Bypass Surgery
Brief Title: Rivaroxaban Effects in Subjects Who Have Undergone Gastric Bypass Surgery
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: PI left the Institution; No replacement PI identified;
Sponsor: State University of New York - Upstate Medical University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SUNYUMU-rivpd-001
Record Dates: First submitted 2014-02-06; First posted 2014-02-07 (Estimated); Last update posted 2016-01-05 (Estimated); Status verified 2015-01

CONDITIONS: Gastric Bypass Status
Keywords: gastric bypass; rivaroxaban; pharmacodynamics
MeSH Terms: interventions — Rivaroxaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- normal subjects (Experimental): A single dose of 10 mg of rivaroxaban will be administered
  Interventions: Drug: rivaroxaban
- Obese non bypassed (Experimental): A single dose of rivaroxaban will be administered
  Interventions: Drug: rivaroxaban
- obese bypassed (Experimental): A single dose of rivaroxaban will be administered
  Interventions: Drug: rivaroxaban
- pre and post bypassed subject (Experimental): A single dose of rivaroxaban will be administered prior to gastric bypass. Subjects will be restudied 12 to 24 weeks following bypass
  Interventions: Drug: rivaroxaban

INTERVENTIONS:
Drug: rivaroxaban — Single dose pharmacodynamic study
  Other Names: Xarelto

SUMMARY:
The investigators are attempting to compare the anticoagulant (blood thinning) effects of a recently FDA approved medication, Rivaroxaban, in people who have undergone gastric bypass surgery to people who have not had this surgery. It is thought that gastric bypass may alter the absorption of this medication, but this has not been previously studied.

The investigators will study the anticoagulant effect of rivaroxaban in healthy volunteers who are in one of four groups

1. Non obese people who have not had a gastric bypass.
2. Obese people who have not had a gastric bypass
3. People who have had a gastric bypass
4. People who are planning to undergo gastric bypass surgery in the near future who are willing to be studied before and after the bypass.

The study will involve taking a single low dose of rivaroxaban and multiple blood samples will be taken over the next 24 hours and the effect of rivaroxaban on blood clotting will be measured using the prothrombin time and an anti-factor Xa assay. The effects of rivaroxaban will be compared between the different groups.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers in one of four groups

  1. Normal weight and not having prior gastric bypass surgery,
  2. Obese and not having prior gastric bypass surgery,
  3. Subjects with prior roux en Y gastric bypass surgery,
  4. Obese and planning to undergo roux en Y gastric bypass

Exclusion Criteria:

* Active renal or liver disease,
* bleeding diathesis,
* concurrent treatment with anticoagulants or aspirin,
* indication for aspirin or anticoagulant treatment,
* gastrointestinal bleeding,
* uncontrolled hypertension,
* active malignancy,
* anemia,
* thrombocytopenia,
* pregnant,
* allergy to rivaroxaban,
* coagulopathy or any other medical condition that would increase risk to the subject

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2014-12; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
median inhibition of factor xa inhibition | 24 hours
  pharmacodynamic

SECONDARY OUTCOMES:
median prolongation of prothrombin time | 24 hours
  pharmacodynamic

CONTACTS AND LOCATIONS:
Overall Officials: Thomas E Coyle, MD, Principal Investigator — State University of New York - Upstate Medical University
Locations (1):
- SUNY Upstate Medical University, Syracuse, New York, United States